CLINICAL TRIAL: NCT02854761
Title: Phase I Safety and Tolerability Study of EF-022 in Adult Subjects With Recurrent Respiratory Papillomatosis
Brief Title: Safety Study of EF-022 in Adults With Recurrent Respiratory Papillomatosis (RRP)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Efranat Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS-102
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Respiratory Papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis

ARMS (2):
- SC administration (Experimental): Subcutaneous (SC) administration of 500 ng of EF-022 (Modified Vitamin D Binding Protein Macrophage Activator) once weekly, for 6 months
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)
- IM administration (Experimental): Intramuscular (IM) adminstration of 500 ng EF-022 (Modified Vitamin D Binding Protein Macrophage Activator) once weekly for 6 months
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)

INTERVENTIONS:
Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)

SUMMARY:
This study evaluates the safety and tolerability of the investigational drug EF-022 in the treatment of adult patients with Recurrent Respiratory Papillomatosis (RRP). Patients will be administered EF-022, either intramuscular or subcutaneous, for a period of 6 months. Preliminary effect of the drug on the disease will be evaluated by following the number and severity of the lesions in the respiratory tract and the effect on voice changes.

DETAILED DESCRIPTION:
The etiology of RRP is associated with local immune suppression at disease-involved sites.

EF-022, a Vitamin D-Binding protein Macrophage Activating Factor, modulates the innate arm of the immune system to alleviate immune suppression. The investigators hypothesize that EF-022 may modulate the immune response in a manner that might slow down or even prevent disease progression.

Adult subjects will be treated weekly with EF-022 for a period of 6 months by either intramuscular or subcutaneous administration.

The primary objective of the study is to evaluate the safety and tolerability of EF-022 administered to adult subjects with recurrent respiratory papillomatosis either IM or SC.

The main response assessment will be performed over the 6 months period by:

* Evaluating lesion size and/or number of disease-involved sites by Coltera-Derkay score
* Assessment of degree of voice disorder using the VHI-10 score
* Symptomatic assessment of dyspnea/stridor

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented diagnosis of recurrent respiratory papillomatosis
2. Patients with measurable disease
3. Patients presenting at least one of the following severity criteria: Derkay score ≥ 8 , Voice handicap index (VHI) ≥11
4. Adult male and female subjects, age of 18 and above (≥18 yrs)
5. Patients with documentation on number of debulking procedures done during past 12 months
6. Estimated expectancy time for next debulking procedure must be at least 3 months.
7. Must be at least 4 weeks (>4 weeks) since last treatment including cytotoxic therapy, biological or immunotherapy, anti-viral therapy, molecularly targeted therapy or steroid treatment.
8. Must be at least 2 weeks (>2weeks) since last NSAID treatment.
9. Must have adequately recovered (to at least Grade 1 level) from adverse effects of prior therapies.
10. Female of child bearing potential must have a negative pregnancy test and must be practicing an effective method of birth control
11. Patients or their guardians must sign an informed consent indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

1. Patient on concurrent steroids or anti-inflammatory non steroid treatment.
2. Active autoimmune disease
3. Known major immunodeficiency
4. Known to be Positive for HIV, Hepatitis B surface antigen, Hepatitis C antibody
5. Have absolute neutrophil counts below 1.5X 10^9/L
6. Hemoglobin below 10.0 g/dL
7. White blood cell counts below 3.5X10^9/L.
8. Granulocytes below 1.5X10^9/L.
9. Have Platelets below 100 X 10^9/L
10. Abnormal renal function with creatinine above 1.5X the upper limit of normal (ULN)
11. Abnormal liver function tests with bilirubin above 1.5X the ULN, AST and ALT above 2.5 X ULN.
12. Patients with active cardiovascular disease under continuous treatment
13. Patients with associated malignancy currently receiving chemotherapy and/or radiation.
14. Female adult patients that are pregnant, nursing or plan to nurse during and up to 12 months of treatment period.
15. Subjects receiving another investigational drug.
16. Patients with concurrent or history of malignancy within 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
CTCAE v.4.03 criteria will constitute the primary safety endpoints to be monitored throughout this study | 6 months